CLINICAL TRIAL: NCT02218385
Title: A Single-arm, Multi-laboratory Clinical Trial of the ForeCYTE Breast Aspirator for Sample Collection, Processing and Cytological Testing of Nipple Aspirate Fluid
Brief Title: ForeCYTE Breast Aspirator for Sample Collection and Cytological Testing of Nipple Aspirate Fluid
Status: Completed | Type: Observational
Sponsor: Atossa Therapeutics, Inc. (Industry)
Collaborators: Quest Diagnostics-Nichols Insitute (Industry); National Reference Laboratory for Breast Health (Unknown); Sound Pathology Associates (Unknown); Puget Sound Institute of Pathology (Other)
Responsible Party: Sponsor
Other Study IDs: GCP003
Record Dates: First submitted 2014-07-30; First posted 2014-08-18 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Breast Neoplasms
Keywords: Nipple Aspirate Fluid; Breast Health Screening; Cytology
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ForeCYTE Breast Aspirator: ForeCYTE Breast Aspirator used for bilateral collection of Nipple Aspirate Fluid (NAF) for cytologic testing
  Interventions: Device: ForeCYTE Breast Aspirator

INTERVENTIONS:
Device: ForeCYTE Breast Aspirator — ForeCYTE Breast Aspirator used for bilateral collection of Nipple Aspirate Fluid (NAF) for cytologic testing

SUMMARY:
The purpose of this study is to measure the performance characteristics for the collection, fixation and transportation of clinical nipple aspirate fluid (NAF) specimens of the ForeCYTE Breast Aspirator across 3 independent labs and the National Reference Laboratory for Breast Health (NRLBH). The study hypothesis is that each lab will have a specimen acceptability rate of at least 90%. If it is assumed that the true level of acceptability testing is approximately 96%, then the lower bound of a one-sided 95% confidence interval is expected to be at least 90%.

DETAILED DESCRIPTION:
A) NAF Collection at physician's office: The Principle Investigator identified and qualified the study subjects. He and the assigned study coordinator from his clinic completed all entries in the Study Case Report Form related to the collection site. He collected the NAF specimens at the Physician Office Collection Sites in accordance with the Instructions for Use.

B) NAF Processing at physician's office: The Principle Investigator's designate processed the NAF specimens for shipment to the selected laboratories in accordance with the Instructions for Use.

C) NAF Transport from physician's office to laboratory: The patient specimen collection membranes were placed in resealable pouches, packed in shipping boxes (provided) and transported by Federal Express to the participating Independent Clinical Laboratories. The Federal Express packaging was pre-labeled for the PI within each of the four laboratories and the specimens were sent in the order in which they were collected to each of the laboratories. Left and right breast specimen from the same subject were sent to the same lab, but in a subject based sequence. The shipments will be shipped serially to lab ABCD, ABCD, ABCD, ABCD, etc. So specimens from subject 1 went to laboratory A, specimens from subject 2 to lab B, specimens from subject 3 to lab C, specimens from subject 4 to lab D, specimens from subject 5 to lab A, etc. The PI completed the Testing Facility Shipping and Receiving Tracking Form for all specimens.

D) NAF Processing at laboratory: The NAF was processed at the clinical cytology laboratories in accordance with the Instructions for Use that accompanied each patient kit.

E) NAF Cytology Classification: A trained, board-certified pathologist read the slides. The data was reported in the Case Report Form according to the format recommended by the College of American Pathologists. The criteria for reading and interpreting the slides are contained in Table 2 and were adapted from King, et al. The laboratory portion of the Case Report Form was completed for each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, female, age 20-75 years, from whom bi-lateral specimens can be obtained.
2. Any woman for whom NAF cytology testing is considered to be beneficial by her physician.
3. Non-lactating and non-pregnant (as documented by date of Last Menstrual Period or post-menopausal).
4. Good general health as determined by medical history, breast disease/cancer history, and clinical breast exam.
5. Willing to give informed consent and follow study procedures as directed.

Exclusion Criteria:

1. Medical condition/psychiatric conditions making subjects a poor candidate for study, as determined by the Principal Investigator.
2. Pregnancy or suspicion of pregnancy.
3. Open cutaneous wounds or atopic dermatitis in the area of the nipple-areolar complex.
4. No or inverted nipple on the breast unfit for fluid collection, or significant prior surgery in the area of the nipple-areolar complex.
5. Participation in an investigational drug or device study less than 30 days prior to enrollment in this study.
6. Pregnancy, childbirth, or lactation less than 90 days prior to enrollment in this study.
7. Acute illness, including taking antibiotics, analgesics, antipyretics and/or cold medications less than 7 days prior to enrollment in this study.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy women, ages 20 to 75 from whom bi-lateral NAF samples can be obtained.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Specimen Acceptance Rate | Within 2 weeks after specimen collection
  A specimen collected, fixated, shipped and received by the reference lab per specification, and rated by the receiving lab as acceptable for cytological testing and interpretation, is deemed acceptable.

SECONDARY OUTCOMES:
Safety / Investigational Device Adverse Effects | Day of specimen collection
  Investigational Device Adverse Effects

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D. Herman, MD, FACOG, Principal Investigator — Elite Women's Health
Locations (1):
- Elite Women's Health, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided